CLINICAL TRIAL: NCT04492085
Title: National Survey of Workplace Violence Against Chinese Physicians of Obstetrics and Gynecology
Brief Title: National Survey of Workplace Violence
Acronym: CMDA-SURVEY1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: CMDA-SURVEY1
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Workplace Violence Against Physicians; National Survey; Obstetrics and Gynecology; China; Random Sample; Questionnaire
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary hospital or clinics
  Interventions: Other: Questionnaire survey
- Secondary hospital
  Interventions: Other: Questionnaire survey
- Tertiary hospital
  Interventions: Other: Questionnaire survey

INTERVENTIONS:
Other: Questionnaire survey — A customized questionnaire will be delivered by the social software WeChat to explore the prevalence, potential reasons and solutions of workplace violence against physicians of obstetrics and gynecology in China

SUMMARY:
China has witnessed a surge in violence against medical personnel, including widely reported incidents of violent abuse, riots, attacks, and protests in hospitals, but little is known about the definite prevalence of workplace violence against physicians of obstetrics and gynecology in China. The aim of this study is to analyze prevalence of workplace violence against physicians of obstetrics and gynecology in China. A customized questionnaire will be delivered by the social software WeChat to the specific hospital which has been randomly sampled, and all physicians of Obstetrics and Gynecology in this hospital will fill the questionnaire anonymously.

A random sampling will be performed in all 32 provinces, municipality or autonomous regions in the mainland of China. It is assumed that acceptable 95% confidence interval is P±4%, and the sample size under the condition of simple random sampling is 600 persons. If the homogeneity is set as 0.15 or 0.2, and each population (unit) has 10 or 15 persons accepting survey, we will achieve a design effect of 2.35 to 3.80. If we choose the design effect of 3, the sample size of every level needs is 1800. Considering 10% population refusing to be surveyed, in all mainland of China, three levels of hospitals will include at least 6000 physicians who accept survey.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old
* Belonging to and registered at specific hospital
* Active employment in obstetrics, reproduction, or gynecology
* Signed an approved informed consents

Exclusion Criteria:

* Not meeting all the inclusion criteria
* Not completing the whole questionnaire

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All physicians of obstetrics and gynecology from the hospitals randomly samples
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-09-27 (Estimated); Study Completion 2020-09-27 (Estimated)

PRIMARY OUTCOMES:
Prevalence of workplace violence in all physicians | In past 12 months
  Percentage of verbal abuse, physical assault and sexual assaults

SECONDARY OUTCOMES:
Potential reasons of workplace violence in all physicians | Two months
  Percentage of different choices of potential reasons in a customized questionnaire
Potential solution of workplace violence in all physicians | Two months
  Percentage of different choices of potential solution in a customized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided